CLINICAL TRIAL: NCT00210795
Title: A Randomized, Double-blind, Placebo-controlled, Study to Assess Changes in Physical Function in Elderly Patients With Anemia of Chronic Disease (ACD) Receiving Epoetin Alfa (PROCRIT�)
Brief Title: A Phase II Study to Assess Changes in Physical Function in Elderly Patients With Chronic Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was stopped due to slow enrollment after enrolling only 12 of 80 patients over 14 months time.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004627
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Aged; Hemoglobins
Keywords: Anemia; Subcutaneous injection; PROCRIT; Erythropoietin; Epoetin Alfa; Hemoglobin Level; Elderly
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to assess changes in physical function in elderly patients (>= 65 years of age) with chronic anemia (Hb <= 11.0 g/dL) due to anemia of unknown cause and receiving weekly subcutaneous doses of Epoetin alfa (PROCRITÂ®) versus placebo

DETAILED DESCRIPTION:
Some elderly patients have a chronic condition that causes anemia (reduction in hemoglobin level, or low red cell count). Anemia occurs commonly with aging and is a frequent medical condition in individuals over the age of 65. Physical performance and function is generally worse in individuals who are anemic. This is a randomized, double-blind, placebo-controlled, multi-center study to assess physical function (to include falls) and fatigue in approximately 80 elderly patients with chronic anemia (anemia present for at least 3 months) and who are receiving weekly PROCRIT. The study will also evaluate hemoglobin levels (oxygen carrying protein in red blood cells), safety, fatigue and cognitive function. The study hypothesis is to demonstrate the study drug will be more effective in treatment of chronic anemia than placebo, resulting in the improvement of physical function and subsequent disabilities, generally well-tolerated. The patients will receive weekly injections of Epoetin alfa (PROCRIT®) or placebo at a starting dose of 10,000 units administered subcutaneously (under the skin).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of chronic anemia defined as a documented Hb value of <= 11.0 g/dL
* No active cancer
* At least 65 years of age with life expectancy of > 6 months
* Community dwelling patients
* Patients with a Short Physical Performance (SPPB) Summary Score of 4-10 at screening and baseline
* Patients with an Mini Mental State Examination (MMSE) score >= 24

Exclusion Criteria:

* Positive stool guaiac test
* Diagnosis of multiple myeloma and/or MGUS
* History of venous thromboembolytic disease
* Previous treatment with Epoetin alfa, Darbepoetin or any form of erythropoietin recently
* Uncontrolled or severe cardiovascular disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-06; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To assess the change in physical function from baseline to end of study as measured by the Short Physical Performance Battery (SPPB) summary score.

SECONDARY OUTCOMES:
To assess efficacy of PROCRIT by achieving a target Hb of 12.5-12.9 g/dL;Change in FACT-An score;Change in Six-Minute Walk Test,Safety (Adverse Event Incidents, Lab Tests and Vital Signs);Cognitive function; Number and type of injuries from falls

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Double-blind, Placebo-controlled, Study to Assess Changes in Physical Function in Elderly Patients with Anemia of Chronic Disease (ACD) Receiving PROCRIT (Epoetin alfa) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=610&filename=CR004627_CSR.pdf